CLINICAL TRIAL: NCT01886326
Title: Peanut Consumption and Human Weight Management
Brief Title: Eating Peanuts for Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Prof. Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0912008773
Record Dates: First submitted 2013-06-19; First posted 2013-06-25 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Obesity; Overweight; Hyperlipidemia
Keywords: Obesity; energy balance; variety; nut intake
MeSH Terms: conditions — Obesity; Overweight; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Consumption of 42 g of salted peanuts (Experimental): Consumption of 42 grams of peanuts daily
  Interventions: Other: Consumption of 42 grams of peanuts daily
- Consumption of 42 g of unsalted peanuts (Experimental): Consumption of 42 grams of peanuts daily
  Interventions: Other: Consumption of 42 grams of peanuts daily
- Consumption of 42 g of spicy peanuts (Experimental): Consumption of 42 grams of peanuts daily
  Interventions: Other: Consumption of 42 grams of peanuts daily
- Consumption of 42 g of honey peanuts (Experimental): Consumption of 42 grams of peanuts daily
  Interventions: Other: Consumption of 42 grams of peanuts daily
- Consumption of 42 g of 3 diff. varieties (Experimental): Consumption of 42 grams of peanuts daily
  Interventions: Other: Consumption of 42 grams of peanuts daily
- Consumption of 42 g of var. of types (Experimental): Consumption of 42 grams of peanuts daily
  Interventions: Other: Consumption of 42 grams of peanuts daily

INTERVENTIONS:
Other: Consumption of 42 grams of peanuts daily — Consumption of the given 42 grams of peanuts daily without instructions for use (i.e. with/without meals, etc.)

SUMMARY:
Evidence is accumulating that peanut consumption confers health benefits, such as reduction of cardiovascular disease risk and possibly diabetes risk (Jenkins et al., 2008; Mattes et al., 2008). However, peanuts are a high fat, energy dense food and concerns about weight gain are widespread. Although research indicates that other characteristics of peanuts offset these properties, and that peanuts may be incorporated into diets without posing a threat to weight gain (Mattes et al., 2008), concern remains among policymakers, healthcare providers, and consumers. Furthermore, worry exists that eating salted peanuts may elevate blood pressure and that eating honey-roasted peanuts make elevate blood sugar. These fears create substantial obstacles to increased peanut consumption.

Recommendations to increase peanut consumption may be made, but if they are not followed, there will be no impact on health. Additional knowledge is needed on: (1) the acceptability of peanuts consumed on a chronic basis, (2) the chronic intake of moderate levels of peanuts and body weight, and 3) the effects of peanuts on blood pressure and blood sugar. The proposed research will examine the acceptability of long-term inclusion of a single form versus varied forms of peanuts in the diet. It is expected that responses will be varied among individuals with different personality characteristics (e.g., prefer sweet versus savory foods, hedonic versus non-hedonic eaters). A better understanding of how different segments of the population choose to include peanuts in their diet and how to optimize long-term consumption should provide insights for better marketing and improved health. Furthermore, it is anticipated that eating salty peanuts will not raise blood pressure and that eating honey-roasted peanuts will not raise blood sugar. Documenting this will add credibility to the evidence that peanuts do not cause weight gain, as well as reinforce recommendations to increase peanut consumption for their health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years of age
* Weight stable (< 3 kg weight change within last 3 months)
* Constant habitual activity patterns (no deviation > 1x/wk at 30 min/session within last 3 months)
* Constant habitual diet patterns within last 3 months
* Willingness to eat all test foods (peanuts daily for 12 weeks)
* No allergy to foods provided in the study (peanuts)
* Not a daily peanut or tree nut consumer
* Not planning to change use of medications known to influence appetite or metabolism
* Not diabetic or hypertensive
* No history of gastrointestinal pathology
* Non-smoker for one year or more

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2010-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in Weight | 2, 4, 6, 8, 10, and 12 weeks
Change in Blood Lipids | 4, 8, and 12 weeks
Change in Blood Pressure | 2, 4, 6, 8, 10, and 12 weeks
Change in Hedonics of peanut consumption | 12 weeks
  Participants will rate their liking of the sample each day using a visual analog scale.
Change in Body Composition | 2, 4, 6, 8, 10, and 12 weeks
Change in Fasting Blood Glucose | 4, 8, and 12 weeks
Change in Cortisol | 4, 8, and 12 weeks
Change in Insulin | 4, 8, and 12 weeks
Change in Pulse | 2, 4, 6, 8, 10, and 12 weeks

SECONDARY OUTCOMES:
Personality Questionnaires | At baseline visit
Flavor attribute liking measures | At baseline
Compliance | 12 weeks
  Participants will self-report compliance to study protocol using record sheets.
Appetitive Ratings | 4, 8, and 12 weeks
  Collected on handheld computer
Consumption Parameters | 12 weeks
  Participants will note if peanuts were eaten as a meal or snack, at what time, and with what other foods daily.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, RD, MPH, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Jones JB, Provost M, Keaver L, Breen C, Ludy MJ, Mattes RD. Effects of daily consumption of one or varied peanut flavors on acceptance and intake. Appetite. 2014 Nov;82:208-12. doi: 10.1016/j.appet.2014.07.023. Epub 2014 Jul 23. PMID 25064672
- [Derived] Jones JB, Provost M, Keaver L, Breen C, Ludy MJ, Mattes RD. A randomized trial on the effects of flavorings on the health benefits of daily peanut consumption. Am J Clin Nutr. 2014 Mar;99(3):490-6. doi: 10.3945/ajcn.113.069401. Epub 2013 Dec 18. PMID 24351876